CLINICAL TRIAL: NCT03015233
Title: Acute Abdominal Pain in Emergency Department: Evaluation of Venous LACtate Value and Strong Ion GAp According to the Stewart Approach as Predictive Factors of Surgical Issue
Brief Title: Acute Abdominal Pain: Evaluation of Lactate Value as Predictive Factor of Surgical Issue
Acronym: GALAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association pour la Formation l'Enseignement et la Recherche du Service de l'Accueil des Urgences (Other)
Responsible Party: Sponsor
Other Study IDs: AFERSAU-2016-01
Record Dates: First submitted 2016-12-23; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Abdomen, Acute; Renal Colic
Keywords: Lactate; Acute Abdominal Pain; Acute Abdomen; Strong Ion Gap; Renal Colic; Emergency Department; Emergency; Surgery; Stewart
MeSH Terms: conditions — Abdomen, Acute; Renal Colic; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Abdominal pain is one of the most common reasons for consultation in Emergency Departments (ED) worldwide. The challenge for physicians is to not misdiagnose a surgical emergency. The actual gold standard for diagnosis is computed tomography (CT). However with this procedure there is high radiation exposure and a risk factor of radiation-induced cancers, therefore alternative diagnostic techniques should be considered. The aim of this study is to evaluate the performance of measuring venous lactate in patients presenting with acute abdominal pain in ED.

In this single-center, prospective, non-interventional study, the diagnostic accuracy of venous lactate in order to detect surgical emergencies is evaluated. The hypothesis made here is that venous lactatemia is a positive predictive factor of surgical emergencies in patients with acute abdominal pain.

DETAILED DESCRIPTION:
Abdominal pain is one of the most common reasons for consultation worldwide in Emergency Departments (ED). The challenge for physicians is to not misdiagnose a surgical emergency. The actual gold standard for diagnosis is computed tomography (CT). However with this procedure there is high radiation exposure and a risk factor of radiation-induced cancers, therefore alternative diagnostic techniques should be considered. The aim of this study is to evaluate the diagnostic performance of measuring venous lactate in patients with acute abdominal pain in ED.

A single-center, prospective, non-interventional study, will be conducted between June 2016 and January 2017 in the university emergency department of Nice, France. Inclusion criteria are patients aged 18 and over, suffering from abdominal pain for seven days or less and requiring a blood test to help with diagnosis.

The primary outcome is to determine if the value of venous lactate is a predictive factor of emergency surgery in patients with acute abdominal pain.

The secondary outcome is to determine if the "strong ion gap", first defined in "The Stewart Approach", is a predictive factor of emergency surgery in patients with acute abdominal pain.

A blood test will be performed when patients are admitted to the ED. Seven days after being admitted to the ED, patients' outcome will be assessed by consulting patients' medical records or by phone call.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patient presenting acute abdominal pain since 7 days or less
* Need of blood sample confirmed by physician
* Affiliation to french social security system
* Informed Consent

Exclusion Criteria:

* Post traumatic abdominal pain / occurrence of abdominal trauma in the 7 days before ED visit
* Patients with cirrhosis classified as Child-Pugh C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting abdominal pain since seven days or less, older than 18 years old, and who need a blood analysis to perform diagnosis after physician's clinical evaluation.
Sampling Method: Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Venous lactate value | At admission of patient in the ED (Day 1) between arrival and up to one hour later
Surgical issue | From Day 1 (D1) to Day 7 (D7)
  The occurence/or not of a surgical outcome in patients with acute abdomen, during the seven days following the ED visit, will be assessed by consulting patients' medical records or by calling them at D7.

SECONDARY OUTCOMES:
Strong ion gap as Stewart approach | At admission of patient in the ED (Day 1) between arrival and up to one hour later
  Strong ion gap (SIG) is a calculated value based on the following equation :
  SIG = (Na+ + K+ + 2xCa2+ + 2xMg2+) - (Cl- - lactate) - HCO3- + albumine x (0.123 x PH - 0.631) + phosphates mesurés x (0.309 x PH - 0.469) All the values are measured on venous samples.

CONTACTS AND LOCATIONS:
Overall Officials: Julie CONTENTI, MD, Study Chair — Association pour la Formation l'Enseignement et la Recherche du Service de l'Accueil des Urgences
Locations (1):
- Nice University Hospital - Pasteur 2, Nice, France, France